CLINICAL TRIAL: NCT04354363
Title: Role of PRP in Intracytoplasmic Sperm Injection in Infertile Women
Brief Title: PRP in Intracytoplasmic Sperm Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ICSI in poor reserve
Record Dates: First submitted 2020-04-17; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PRP (Active Comparator): women who will receive PRP before ICSI
  Interventions: Other: Platelet rich plasma
- No PRP (No Intervention): women who willnot receive PRP before ICSI

INTERVENTIONS:
Other: Platelet rich plasma — Giving women PRP before ICSI
  Arms: PRP

SUMMARY:
Infertility is a major problem nowadays

DETAILED DESCRIPTION:
ovarian and uterine factor of infertility are very hard to treat

ELIGIBILITY:
Inclusion Criteria:

* women with primary infertility

Exclusion Criteria:

* women with unexplained infertility

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — women with infertility
Enrollment: 60 (Estimated)
Dates: Start 2020-04-22 (Estimated); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
The number of women wo will have chemical pregnancy | within 3 months
  how many women will have chemical pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Study Chair — Algezeera hospitaland National Research Centre ,Egypt
Locations (1):
- Algazeerah, Giza, Egypt